CLINICAL TRIAL: NCT02211352
Title: Randomized Control Clinical Trial for Effect of Korean Red Ginseng on Central Blood Pressure in Patient With Essential Hypertension
Brief Title: Effect of Korean Red Ginseng on Central Blood Pressure in Patient With Essential Hypertension
Acronym: KRGCBP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daegu Catholic University Medical Center (Other)
Collaborators: The Korean Society of Ginseng (Other)
Responsible Party: Principal Investigator, Jin Bae Lee, Associate professor, Daegu Catholic University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: GS302-100; GS302-100 (Other Grant/Funding Number: GS302-100)
Record Dates: First submitted 2013-05-01; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension
Keywords: blood pressure, ginseng
MeSH Terms: conditions — Hypertension | interventions — Asian ginseng; Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active(Korean Red Ginseng) first group: (Active Comparator): Korean Red Ginseng Capsules 2g,daily, 8 week and than crossover to placebo capsules(2g), daily 8week
  Interventions: Drug: Korean Red Ginseng Capsules
- Placebo capsules (Placebo Comparator): placebo Capsules(2g),daily, 8 week and than crossover to Korean Red Ginseng capsules(2g), daily 8week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Korean Red Ginseng Capsules — Korean Red Ginseng Capsules 2mg,daily, 8 week and than crossover to placebo capsules(2g), daily 8week
  Other Names: Korean Red Ginseng (KRG) Capsule was manufactured; from roots of a 6-year-old Panax ginseng Meyer.
  Arms: Active(Korean Red Ginseng) first group:
Drug: Placebo — Korean Red Ginseng Capsules 2mg,daily, 8 week and than crossover to placebo capsules(2g), daily 8week
  Other Names: Placebo of Kerea Red Ginseng(KRG) Capsule
  Arms: Placebo capsules

SUMMARY:
The purpose of this study is to determine Korean red ginseng (KRG)treatment could decrease central blood pressure in subjects with hypertension.

DETAILED DESCRIPTION:
Participants with hypertension who were treated with antihypertensive agents were randomly assigned to an active (KRG 2 g/day) or a placebo treatment group in a double-blind cross over manner.

Participants were not allowed to change their antihypertensive medications except safety issue. Brachial systolic BP (SBP), diastolic BP (DBP), Central SBP and DBP will measured at baseline,at 2 and 4 months.

Efficacy and safety data will be monitored by Daegu Catholic University Medical Center Institutional Review Board and reported to the Korean Ginseng Society.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension
* diastolic blood pressure 100 mmHg or less and systolic blood pressure 160 mmHg or less

Exclusion Criteria:

* Secondary hypertension
* Serum creatinin above 1.5 mg/dL
* aspartate aminotransferase(AST) and alanine aminotransferaseALT above two times upper normal limits
* Uncontrolled diabetes (Hb A1c < 9%)
* Acute myocardial infarction or coronary artery disease intervention within six months
* Moderate to severe congestive heart failure
* HIV positive
* Immunocompromized host
* Allergy to Korean red ginseng
* Pregnancy or plan to pregnancy
* Alcohol or drug abuse
* Attend to other clinical trial within 12 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
central blood pressure change after treatment of Korea Red Ginseng | baseline, 8 weeks and 16 weeks after treatment

SECONDARY OUTCOMES:
brachial systolic and diastolic blood pressure | baseline, 8 week, 16 week.
Augumentation index | baseline, 8 week, 16 week.
ESR(erythrocyte sedmentation rate) | baseline, 8 week, 16 week.
CRP(C-reactive protein) | baseline, 8 week, 16 week.

OTHER OUTCOMES:
AST(Aspartate Aminotransferase) | baseline, 8 week, 16 week
Number of participants with adverse events | baseline, 8 week, 16 week
fasting blood glucose | baseline, 8 week, 16 week
Hb A1c(Hemoglobin A1c) | baseline, 8 week, 16 week

CONTACTS AND LOCATIONS:
Overall Officials: Jin Bae Lee, MD, PhD, Principal Investigator — Daegu Catholic University Medical Center
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea